CLINICAL TRIAL: NCT00361751
Title: Phase 2 Trial to Examine the Metabolic Effects of Fenofibrate in Burned Patients
Brief Title: Substrate Cycling in Energy Metabolism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Shriners Hospitals for Children (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DK34817 (completed)
Record Dates: First submitted 2006-08-07; First posted 2006-08-09 (Estimated); Last update posted 2010-02-15 (Estimated); Status verified 2010-02

CONDITIONS: Burns; Insulin Resistance
Keywords: Glucose metabolism; Fat Metabolism; Insulin Resistance; Protein Metabolism; Tracer Methodology
MeSH Terms: conditions — Burns; Insulin Resistance | interventions — Fenofibrate

INTERVENTIONS:
Drug: fenofibrate

SUMMARY:
Insulin resistance and hyperglycemia contribute to negative outcomes in burned patients. We will assess insulin sensitivity in traditional terms of glucose metabolism, and with regard to the responsiveness of both muscle and liver protein metabolism, in severely burned patients. Plasma free fatty acid (FFA) and tissue TG levels will be manipulated via inhibition of peripheral lipolysis with nicotinic acid or activation of plasma lipoprotein lipase activity with heparin, stimulation of tissue fatty acid oxidation and thus reduction of tissue TG with the peroxisome proliferate-activated receptor (PPAR) alpha agonist fenofibrate. Methodological approaches will include stable isotope tracer techniques to quantify kinetic responses of protein, glucose and lipid metabolism in vivo, quantification of intracellular stores of TG and glycogen by means of magnetic resonance spectroscopy (MRS), as well as quantitative analysis of tissue levels of active products of fatty acids, key intermediates of the insulin signaling pathway, glycogen, the enzyme activities of citrate synthase and glycogen synthase and the activity of the muscle mitochondria. These studies will clarify the physiological and clinical significance of the alterations of tissue lipid metabolism that occur after burn injury, thereby forming the basis for new therapeutic approaches not only in this specific clinical condition but in other clinical circumstances in which hepatic and/or muscle TG is elevated.

We will investigate the general hypothesis that the accumulation of intracellular TG in liver and muscle either directly causes insulin resistance in those tissues or serves as an indictor of the intracellular accumulation of active fatty acid products, such as fatty acyl CoA and diacylglycerol, which in turn disrupt insulin action.

The following specific hypotheses will be investigated:

1. Intracellular TG is elevated in both muscle and liver in severely burned patients. The reduction of the fat in the liver and the insulin resistance will improve clinical outcomes, glucose and protein metabolism.
2. The insulin signaling pathway, as reflected by phosphoinositol-3-kinase (PI3K) and PKC activity, is impaired in tissues with elevated TG.
3. Fatty acids, or their active intracellular products, are the direct inhibitors of insulin action, rather than the tissue TG itself.

DETAILED DESCRIPTION:
We will study patients with severe burns, defined as 2nd or 3rd degree burn covering >40% of total body surface area (TBSA). We propose to study burned children from Shriners Burns Hospital. The Shriners census is such that approximately 50 children with severe burns are treated every year. We will study patients immediately prior to their third surgical procedure, approximately 12-15 days after injury. One half of the patients will be given fenofibrate (5 mg/kg/day) daily delivered through feeding tube from the time of consent following admission until 12-14 days post-burn. This length of time after injury will ensure that untreated patients will have a large accumulation of hepatic TG. Because the "control" group of patients will have elevated liver TGs, the "experimental" group will have their hepatic TGs lowered by fenofibrate. By studying the patients the day before the operations, it will be possible to remove the staples used in skin grafting without risk of loss of adhesion of the graph, thereby ensuring safety in the MRS. Femoral line inserted for the surgery can also be utilized, and all patient generally receive a full transfusion during surgeries, minimizing any study related blood loss. In addition to the liver, we will study the muscle in burn patients. Patients will be studied during brief fasted state. The will be fasted four hours prior to the study and then through out the study. Their TPN will be immediately reconnected following the study. The surgical team at the Shrine places 3Fr, 8 cm polyethylene catheters (Cook, Inc., Bloomington, IN) into the femoral vein and femoral artery under local anesthesia the day before surgery. Both femoral catheters will be used for blood sampling, while the femoral arterial catheter will also used for indocyanine green infusion for the determination of leg blood flow. Systemic concentration of indocyanine green will be measured from a central vein, as standard procedure has a multi-lumen subclavian line in all patients. Patency of all catheters is maintained by saline infusion.

Patients will be infused with stable (non-radioactive) isotope tracers of glucose, phenylalanine and palmitate for up to 8 hours. After 4 hours, without interruption of the tracer infusion, an infusion of insulin will be started and maintained at the rate of 1.5 mU/kg•min for the final 4 h. Blood glucose concentrations will be measured throughout the insulin infusion and glucose infused as necessary to maintain the basal plasma glucose concentration.

A biopsy of the quadriceps will be obtained with a Bergstrom needle at the beginning of the study, 4 h (immediately before the insulin infusion) and at the end of the 4 h insulin infusion. We will use the A-V balance technique to address the relation between tissue fatty acid and TG metabolism and the insulin responsiveness of glucose uptake and myofibrillar and mitochondrial protein synthesis and net protein balance.

b. Subjects Patients are admitted to the burn unit within 48 h of injury. Fluid resuscitation is provided as previously described (94). Within 48 h of admission, the burn wound is excised and subsequently grafted by autograft or cadaveric allograft. Patients typically return to the operating room for reharvesting of donor sites every five to seven days. The experiments proposed here will be performed the day prior to the third surgery at day 12-15, as femoral catheters are normally inserted at the time for access during surgery. Enteral feeding with Vivonex TEN (Sandoz Nutrition Corp, Minneapolis, MN) is started within 24h of admission and continued until the patient is capable of food by mouth. All patients will be eligible for the study unless one of the exclusion criterion listed below apply.

c. Procedures From day 1 to day 22 patients will be maintained on enteral feeding of a high carbohydrate/amino acid mixture (Vivonex, Novartis, Minneapolis, MN). Vivonex contains 300 kcal/serving in the following caloric breakdown: 82.3% carbohydrate, 15% protein, 2.7% fat (linoleic acid). Patients will be given 25 kcal/kg of Vivonex plus an additional 45 kcal/kg for each percentage point of total body surface area burned. One half of the patients will be given fenofibrate (5 mg/kg/day - maximum daily dose) from the time of the first tracer study until the time of the second tracer study.

The tracer study subjects can commence once catheters in the femoral artery and vein have been placed by the surgical team, if necessary, since the majority of patients wil have pre-existing lines placed for clinical reasons. The catheters will be used for sampling and in a peripheral vein for infusing, as in our previous studies (e.g., 4). Enteral administration of a mixture of carbohydrate and amino acids (Vivonex) will be stopped four hours prior to the study, and will be started immediately following the study.

On the day after the tracer infusion the amount of liver and muscle TG and liver glycogen will be determined by MRS. After metal staples are removed, patients will be transported to the clinical MRS facilities at UTMB Dept. of Radiology, where measurements will be performed (see below for details), After obtaining baseline samples, tracer infusions will be started as described in Figure 2. Half the patients with high tissue TG will be given nicotinic acid (500 mg orally) at the start of period 2 to lower FFA levels acutely. In the group given fenofibrate (200 mg/d) or propranolol 0.5mg/kg every 6 hours to lower FFA, half will be infused with heparin (0.5 U/kg•min, 2.8 U/ kg prime IV) at a dose sufficient to activate lipoprotein lipase, thereby elevating plasma FFA, while not affecting blood coagulation. After baseline blood samples from the femoral artery, femoral vein, and peripheral vein are collected, an 8 hour continuous infusion of primed-constant infusions of 6,6-d2-glucose (0.08 mg/kg•min, prime = 6.8 mg/kg) and d5-phenylalanine (0.20 µmol/kg•min, prime = 8.0 µmol/kg) will be given in order to quantify hepatic glucose production and protein synthetic rates, respectively. In addition, 2 hours into the protocol, U-13C16-palmitate (0.16 µmol/kg per minute) will be started with NaH13CO3 prime (150 µmol/kg) in order to quantify hepatic fatty acid uptake and oxidation. These tracer infusions will also be maintained throughout the 8 hour tracer study. Blood samples (2- 12 ml) will be taken from the artery, femoral vein and peripheral vein simultaneously at 120, 180, 210, 225 and 240 minutes (see Appendix 2 for full timeline). Muscle tissue biopsies will be obtained at the start of period 1, and at 4 hours of period 1 to measure protein kinetics and also determine biochemical parameters. Then, period 2 will start. At the start of period 2, a primed, constant infusion of 15N-phenylalanine will be started and maintained throughout period 2. The different tracer of phenylalanine will be used to quantify the plasma protein synthetic rates using the same tracer protocol as in period 1. We have previously shown that the two phenylalanine tracers yield the same results (70). The tracer technique will enable us to measure the primary endpoints of insulin responsiveness of the liver, i.e., endogenous glucose production and synthetic rates of albumin and fibrinogen. At 4 hours, hyperinsulinemia will be initiated by the infusion of insulin at the rate of 1.5 mu/kg•min, which will result in circulating levels of approximately 200 uU/ml (5). This rate of infusion was based on our previous experience with insulin infusion in burned patients (e.g., 1-5). We anticipate a considerable variation in the baseline insulin concentrations, such that if a low rate of infusion were to be used, the resulting "hyperinsulinemia" in some patients would likely be below the baseline concentration in others. Consequently, we have chosen a rate of infusion that will result in a clear-cut difference between the baseline and "hyperinsulinemic" values. Further, although during the insulin infusion we anticipate that insulin concentrations will also be variable, our endpoints will be assessed in terms of the magnitude of change from the baseline value in each subject. This statistical approach should minimize concern regarding subject variability. The dosage was selected because we have previously shown that protein metabolism is responsive to this rate of infusion (5), but that it is below the maximally-effective dose (4). Blood glucose concentration will be monitored throughout the second period, and glucose will be infused (if necessary) to maintain glucose concentrations at the baseline level. Since the baseline concentrations of glucose will vary, this means that during hyperinsulinemia the glucose concentrations will likely differ between subjects, but we have selected this approach because in this way only the insulin concentration will differ between periods 1 and 2, thereby simplifying interpretation of the changes in substrate and protein kinetics from period 1 to 2. The sampling schedule will be the same as in period 1, including the timing of the biopsy (i.e., at 4 h of period 2).

Leg blood flow will be measured by indocyanine green infusion, ad described previously (14). Whole-body indirect calorimetry will be performed to quantify whole-body carbohydrate and fat oxidation.

ELIGIBILITY:
Inclusion Criteria:

We will study male and female burned patients from 20 KG (based on blood requirement) in weight. Patients will be studied between days 12-15 after the initial surgery and will have burns constituting >40% of the body surface. Volunteers will be determined as healthy utilizing history, physical examination and screening laboratory values assessing liver and renal function, coagulation and platelet function.

Exclusion Criteria:

1.Sulfide or iodide allergies 2.Respiratory Insufficiency 3.Multiple Fractures 4.History of Cancer in the last 5 years 5.Diabetes Mellitus 6.Bilirubin >3.0 mg/dl 7.Associated head injuries requiring specific therapy 8.Associated injuries to chest or abdomen requiring surgery 9.Serum creatine > 3.0 mg/dl after fluid resuscitation 10.Receipt of any experimental drug other than ones supplied with two months of this study 11.Any metal in body including rods, neurofibrilators, pacemakers, etc. 12.Orthopedic casting which would prevent placement in MRI 13.Hepatitis 14.Abnormal EKG 17. Bruits over the femoral artery 18. Electrical burn 19. Patients unable to lie still without heavy sedation will not be used for the MRS portion of the study.

-

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40
Dates: Start 2003-05; Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Daily Plasma Glucose
Insulin stimulated glucose uptake
Hepatic fat concentration
Muscle fat concentrations and species

SECONDARY OUTCOMES:
Muscle insulin signalling
Muscle mitochondrial function
Muscle mitochondrial enzyme activity
Hepatic protein production
Muscle protein balance
Whole Body palmitate oxidation
FFA release/balance
Resting Energy Expenditure
Body Mass Composition

CONTACTS AND LOCATIONS:
Overall Officials: Robert R Wolfe, PhD, Principal Investigator — UTMB/University of Arkansas
Locations (1):
- Shriners Hospital for CHildren, Galveston, Texas, United States

REFERENCES:
- [Derived] Cree MG, Zwetsloot JJ, Herndon DN, Qian T, Morio B, Fram R, Sanford AP, Aarsland A, Wolfe RR. Insulin sensitivity and mitochondrial function are improved in children with burn injury during a randomized controlled trial of fenofibrate. Ann Surg. 2007 Feb;245(2):214-21. doi: 10.1097/01.sla.0000250409.51289.ca. PMID 17245174